CLINICAL TRIAL: NCT01025635
Title: Randomized, Double-blind, Vehicle-controlled, Multicenter, Parallel-group Study to Investigate Safety and Efficacy of Azelaic Acid Foam, 15% Topically Applied Twice Daily in Subjects With Papulopustular Rosacea
Brief Title: Safety and Efficacy of Azelaic Acid Foam, 15% in Papulopustular Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14955; 1403120 (Other: Company internal)
Record Dates: First submitted 2009-11-26; First posted 2009-12-03 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2014-04

CONDITIONS: Papulopustular Rosacea
Keywords: rosacea; papulopustular; azelaic acid; foam
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azelaic acid foam, 15% (BAY39-6251) (Experimental): Participants received azelaic acid foam, 15% topically twice daily for 12 weeks
  Interventions: Drug: Azelaic acid foam 15%
- Vehicle foam (Placebo Comparator): Participants received vehicle foam topically twice daily for 12 weeks
  Interventions: Drug: Vehicle foam

INTERVENTIONS:
Drug: Azelaic acid foam 15% — Applied topically twice daily for 12 weeks
  Arms: Azelaic acid foam, 15% (BAY39-6251)
Drug: Vehicle foam — Applied topically twice daily for 12 weeks
  Arms: Vehicle foam

SUMMARY:
This study will investigate the safety and efficacy of a new formulation of an existing medication for the treatment of papulopustular rosacea. The study will test the active ingredient plus foam against foam alone.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Diagnosis of papulopustular rosacea (IGA score of moderate or severe) with a minimum of 12 and maximum of 50 inflammatory lesions (papules and/or pustules) and persistent erythema with or without telangiectasia
* Free of any clinically significant disease which could interfere with the study
* Willingness to follow all study procedures
* Male or female patient at least 18 years of age

Exclusion Criteria:

* Subjects known to be non-responders to azelaic acid
* Presence of dermatoses that might interfere with the rosacea diagnosis or the evaluation of treatment results
* Ocular rosacea, phymatous rosacea
* Any condition or therapy that in the opinion of the investigator may pose a risk to the patient of interfere with any evaluation in the study
* Facial laser surgery in the 6 weeks prior to the study
* Topical or systemic use of prescription or non-prescription medications to treat rosacea
* Use of any agent other than the investigational drugs to treat rosacea during the study
* Expected use or change in dose in the 90 days prior to the study of beta-blockers, vasodilators, NSAIDs, hormonal treatment or drugs causing acneiform eruptions
* Known hypersensitivity to any ingredients of the investigational product formulation
* Alcohol or drug abuse
* Incapability of giving fully informed consent
* Subject is dependent person, i.e., a relative/family member of the investigator and/or is a member of the investigator's staff
* Participation in another clinical research study within the last 4 weeks before randomization in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2009-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (19):
- United States (19):
  - Birmingham, Alabama
  - Fremont, California
  - Santa Monica, California
  - Miami, Florida
  - Miramar, Florida
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - High Point, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Portland, Oregon
  - Johnston, Rhode Island
  - Simpsonville, South Carolina
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Plano, Texas
  - Salt Lake City, Utah
  - Madison, Wisconsin

REFERENCES:
- [Background] Draelos ZD, Elewski B, Staedtler G, Havlickova B. Azelaic acid foam 15% in the treatment of papulopustular rosacea: a randomized, double-blind, vehicle-controlled study. Cutis. 2013 Dec;92(6):306-17. PMID 24416747

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Started | 198 | 203
Completed | 175 | 178
Not Completed | 23 | 25
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Protocol Violation | 4 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 9 | 13
Not completed — Reason not known | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam | Total
Number analyzed (Participants) | 198 | 203 | 401
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.1 (12.23) | 48.9 (11.65) | 48.5 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 143 | 298
  Male | 43 | 60 | 103
Previous duration of rosacea [Mean (Standard Deviation); unit: Months] | 121.4 (113.38) | 126.3 (103.81) | 123.8 (108.53)
Investigator's Global Assessment (IGA) score at Baseline [Mean (Standard Deviation); unit: Scores on a scale] — IGA categories: 0 - Clear; 1 - Minimal; 2 - Mild; 4 - Moderate; 6 - Severe / Therapeutic success is defined as an IGA score of clear or minimal (0 to 1).
  Scores on a scale | 4.3 (0.68) | 4.1 (0.51) | 4.2 (0.60)
Number of inflammatory lesions per participant at Baseline [Mean (Standard Deviation); unit: Inflammatory lesions] | 21.6 (9.91) | 20.4 (8.83) | 21.0 (9.38)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Based Therapeutic Success at End of Treatment (LOCF: Last Observation Carried Forward)
Description: The IGA is a static evaluation of the overall severity of papulopustular rosacea at a given time. It consists of 5 scores ranging from clear to severe papulopustular rosacea and allows rapid overall evaluation of disease severity: 1) Clear: virtually no rosacea, ie, no papules and/or pustules; no erythema; 2) Minimal: rare papules and/or pustules; residual to mild erythema; 3) Mild: few papules and/or pustules; mild erythema; 4) Moderate: pronounced number of papules and/or pustules; moderate erythema; 5) Severe: numerous papules and/or pustules, occasionally with confluent areas of inflamed lesions; moderate to severe erythema. Therapeutic success is defined as an IGA score of clear or minimal.
Time Frame: At End of treatment (up to 12 weeks) (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 198 | 203
Percentage of participants | 43.4 | 32.5
Statistical Analysis 1: Comparison: Azelaic Acid Foam, 15% (BAY39-6251) vs Vehicle Foam; Test type: Superiority or Other; p = 0.017, Cochran-Mantel-Haenszel; study center adjusted

2. Primary Outcome: Nominal Change From Baseline in Inflammatory Lesion (IL) Count (Sum of Papules and Pustules) Per Participant at End of Treatment (LOCF)
Time Frame: Baseline and End of treatment (up to 12 weeks) (LOCF)
Measure: Mean (Standard Deviation); unit: Inflammatory lesions
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 198 | 203
Inflammatory lesions | -13.4 (10.39) | -9.5 (9.73)
Statistical Analysis 1: Comparison: Azelaic Acid Foam, 15% (BAY39-6251) vs Vehicle Foam; Test type: Superiority or Other; p < 0.001, ANCOVA; with factors treatment group, study center, and baseline lesion count as covariate

3. Secondary Outcome: Percent Change From Baseline in IL Count (Sum of Papules and Pustules) Per Participant at End of Treatment (LOCF)
Time Frame: At End of treatment (up to 12 weeks) (LOCF)
Measure: Mean (Standard Deviation); unit: Percentage of Inflammatory lesions
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 198 | 203
Percentage of Inflammatory lesions | -62.5 (35.66) | -47.8 (41.28)

4. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Based Patient Response at End of Treatment (LOCF)
Description: The IGA is a static evaluation of the overall severity of papulopustular rosacea at a given time. It consists of 5 scores ranging from clear to severe papulopustular rosacea and allows rapid overall evaluation of disease severity: 1) Clear: virtually no rosacea, ie, no papules and/or pustules; no erythema; 2) Minimal: rare papules and/or pustules; residual to mild erythema; 3) Mild: few papules and/or pustules; mild erythema; 4) Moderate: pronounced number of papules and/or pustules; moderate erythema; 5) Severe: numerous papules and/or pustules, occasionally with confluent areas of inflamed lesions; moderate to severe erythema. Subjects achieving a clear, minimal, or mild IGA at the end of treatment were considered as 'responder'. Subjects with an IGA of moderate or severe at the end of treatment were considered as 'non-responder'. Subjects who prematurely withdraw from study treatment because of lack of efficacy were coded as 'non-responders'.
Time Frame: At End of treatment (up to 12 weeks) (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 198 | 203
Percentage of participants | 69.2 | 57.6

ADVERSE EVENTS:
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Serious Adverse Events (participants affected / at risk) | 1/198 | 3/203
Other Adverse Events (participants affected / at risk) | 68/198 | 48/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azelaic Acid Foam, 15% (BAY39-6251) (N=198) | Vehicle Foam (N=203)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azelaic Acid Foam, 15% (BAY39-6251) (N=198) | Vehicle Foam (N=203)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 0 (0) | 1 (1)
Application site pain (General disorders) | 9 (9) | 3 (4)
Application site pruritus (General disorders) | 3 (3) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2)
Cyst (General disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 7 (7) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1)
Tenderness (General disorders) | 1 (2) | 0 (0)
Application site dryness (General disorders) | 0 (0) | 1 (1)
Application site paraesthesia (General disorders) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (7) | 6 (6)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Whiplash injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Burning sensation (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 9 (21) | 2 (3)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dental care (Surgical and medical procedures) | 1 (1) | 0 (0)
Mammoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the results of Study only after review, comment and approval by Intendis. At least sixty (60) days prior to submitting a manuscript to a publisher or other outside persons (i.e., reviewer(s)) or prior to any public presentation), a copy of the manuscript or presentation will be provided to Intendis by the Investigator for review and comment. No publication of confidential information shall be made without Intendis' prior written consent.